CLINICAL TRIAL: NCT01339104
Title: An Open-label, Non-randomized Phase I Study of Regorafenib (BAY73-4506) to Evaluate Cardiovascular Safety Parameters, Tolerability, Pharmacokinetics, and Anti-tumor Activity in Patients With Advanced Solid Tumors
Brief Title: Open Label Regorafenib Study to Evaluate Cardiovascular Safety Parameters, Tolerability, and Anti-tumor Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14814
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Neoplasms
Keywords: Cardiovascular safety
MeSH Terms: conditions — Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regorafenib (Experimental)
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — All subjects will receive regorafenib administered from Day 1 -21 at a dose of 160 mg od (4 x 40 mg tablets) followed by a 7 days break in repeating cycles of 28 days. The drug is to be taken in the morning with approximately 240 mL of water after having a low fat breakfast. Holter ECGs with triplicate measurements will automatically be obtained at specified timepoints over 24 hours on days -1 and Cycle 1, Day 21. PK samples will be drawn on Cycle 1, Day 21. PK timepoints are time-matched with Holter ECG timepoints. 24 hour urine will be collected beginning on Cycle 1, Day 21. MUGA scans will be done at screening, Cycle 2 Day 21 (after 42 doses of BAY73-4506), then every 3 cycles starting in Cycle 5, and at end of treatment.

SUMMARY:
Open label Phase I study of Regorafenib to evaluate cardiovascular safety, tolerability and anti-tumor activity in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects >/= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
* Adequate bone marrow, liver, and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to dosing:

  * Hemoglobin (Hb) >/= 9.0 g/dL, Absolute neutrophil count (ANC) >/= 1500/mm³, Platelet >/= 100,000/mm³, Total bilirubin </= 1.5 times upper limit of normal (ULN), Alkaline phosphatase </= 4 x ULN
  * Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) </= 2.5 times ULN (</= 5.0 x ULN for subjects with liver involvement of their cancer), International Normalized Ratio (INR) or Partial Thromboplastin Time (PTT) < 1.5 x ULN, Serum creatinine </= 1.5 times ULN and glomerular filtration rate (GFR) >/= 30 ml/min/1.73 m² according to the MDRD (Modified Diet in Renal Disease) abbreviated formula, Lipase </= 1.5 x ULN
  * Left Ventricular Ejection Fraction (LVEF) >/= 50 % as assessed at the Baseline Multigated Acquisition (MUGA) scan
  * QTc (Q-T corrected) </= 470 msec at Screening
* Having advanced, refractory disease
* Life expectancy of at least 3 months
* Recovery from any previous drug/procedure-related toxicity to Common Toxicological Criteria (CTC) Grade 0 or 1 levels (except alopecia), or to baseline preceding the prior treatment.

Exclusion Criteria:

* History of cardiac disease: congestive heart failure > New York Heart Association (NYHA) Class II; active coronary artery disease (unstable angina [anginal symptoms at rest] or new-onset angina [began within the last 3 months] or myocardial infarction within the past 6 months).
* Uncontrolled hypertension (failure of diastolic blood pressure to fall below 90 mmHg, despite the use of >/= 3 antihypertensive drugs or systolic blood pressure greater than 150 mmHg)
* History of or known human immunodeficiency virus (HIV) infection or active hepatitis B or C.
* Subjects with serious non-healing wound, ulcer, or bone fracture
* Subjects with arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within the 6 months before start of study medication
* Persistent proteinuria of CTC Grade 3 or higher (> 3.5 g/24 hours, measured by urine protein/creatinine ratio on a random urine sample)
* Symptomatic metastatic brain or meningeal tumors unless the subject is > 6 months from definitive therapy, has no evidence of tumor growth on an imaging study within 2 weeks prior to study entry, and is clinically stable with respect to the tumor at the time of study entry
* Clinically significant bleeding (CTC AE Grade 3 or higher) within 30 days before start of study medication.
* Subjects with seizure disorder requiring anticonvulsant medication
* History of organ allograft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Effect of regorafenib on cardiovascular safety parameters measured by change in QT\QTc on the ECG in patients with advanced solid tumors | After 8 weeks
Effect on Left Ventricular Ejection Fraction (LVEF) | 12 weeks post Cycle 1

SECONDARY OUTCOMES:
Decrease in tumor size based on investigator assessed RECIST criteria | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- United States (6):
  - Aurora, Colorado
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee
  - Seattle, Washington

REFERENCES:
- [Derived] Jones RL, Bendell JC, Smith DC, Diefenbach K, Lettieri J, Boix O, Lockhart AC, O'Bryant C, Moore KN. A phase I open-label trial evaluating the cardiovascular safety of regorafenib in patients with advanced cancer. Cancer Chemother Pharmacol. 2015 Oct;76(4):777-84. doi: 10.1007/s00280-015-2827-3. Epub 2015 Aug 18. PMID 26281907